CLINICAL TRIAL: NCT01705275
Title: A Randomised, Double-blind, Placebo-controlled, Two-period Crossover Study to Investigate the Effect of ONO-8539 on Acid-induced Oesophageal Hypersensitivity in Healthy Male Adult Volunteers
Brief Title: A Study to Investigate the Effect of ONO-8539 on Acid-Induced Oesophageal Hypersensitivity in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-8539POE012
Record Dates: First submitted 2012-08-03; First posted 2012-10-12 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2012-10

CONDITIONS: Acid Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ONO-8539

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONO-8539 BID (Experimental): ONO-8539
  Interventions: Drug: ONO-8539
- Placebo BID (Placebo Comparator): 0mg
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ONO-8539 — ONO-8539
  Other Names: ONO-8539 acid hypersensitivity
  Arms: ONO-8539 BID
Other: Placebo — Identical to ONO-8539 tablet but without active ingedient
  Other Names: 0mg ONO-8539
  Arms: Placebo BID

SUMMARY:
A study to investigate the efficacy of ONO-8539 on acid-induced oesophageal hypersensitivity in healthy male adult volunteers.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, two-period crossover study, to investigate the efficacy of ONO-8539 on acid-induced oesophageal hypersensitivity in healthy male adult volunteers. Each subject will be randomised to ONO-8539 or placebo twice daily in the first treatment period and the alternate treatment in the second treatment period. Dosing in each period will be for 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects, aged 18-45 years inclusive, will be entered into this study.

Exclusion Criteria:

* Subjects will be excluded if they have a motility disorder, are not able to tolerate study procedures or have had GI surgery or have a condition that would affect the study results.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the change from baseline in pain threshold in the proximal oesophagus following electrical stimulation after oesophageal acid infusion. | 15 days

SECONDARY OUTCOMES:
Area under the Curve (AUC) of the change from baseline in pain threshold in the distal oesophagus following electrical stimulation after oesophageal acid infusion | 15 days
Maximum change from baseline in pain threshold in the proximal and distal oesophagus following electrical stimulation after oesophageal acid infusion. | 15 days
Change in absolute pain threshold from baseline in the proximal and distal oesophagus and somatic control following electrical stimulation after oesophageal acid infusion at each time point. | 15 Days
Change from baseline at each time point in subject reported pain following electrical stimulation after oesophageal acid infusion using the short-form McGill pain questionnaire (SF-MPQ). | 15 Days
Relationship between the pharmacokinetics of ONO-8539 and change from baseline in pain threshold in the proximal oesophagus following electrical stimulation after oesophageal acid infusion. | 15 Days
Relationship between State Trait Anxiety Inventory (STAI)-state score and change from baseline in pain threshold in the proximal oesophagus following electrical stimulation after oesophageal acid infusion. | 15 Days
Safety and tolerability: adverse events, physical examination, body weight, vital signs, 12-lead Electrocardiogram (ECG) and safety laboratory evaluations. | 15 Days
The maximum observed plasma concentrations (Cmax), time to reach Cmax (Tmax), area under the curve (AUC), and trough concentration of ONO-8539 prior to dosing. | 15 Days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Clinical Department, Ono Pharmaceutical Co. Ltd
Locations (1):
- London Clinical site Recruiting, London, London, United Kingdom